CLINICAL TRIAL: NCT05562739
Title: A Randomized, Double-blinded, Placebo-controlled, Parallel Pilot Study, to Assess the Effect of a Postbiotic Blend on Symptoms of Anxiety in Healthy Adults with Self-reported Mild to Moderate Anxiety
Brief Title: Pilot Study to Assess the Effect of a Postbiotic Blend on Moderate Self-reported Anxiety
Acronym: Anx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Archer-Daniels-Midland Company (Industry)
Collaborators: Atlantia Food Clinical Trials (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTB2022TN105P2
Record Dates: First submitted 2022-09-28; First posted 2022-10-03 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Anxiety
Keywords: probiotic; microbiome; postbiotic
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: This is part 2 of a study with the participants being recruited from "Placebo non-responders" in Part 1 of the study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active (Experimental): Arm receiving investigational product (postbiotic)
  Interventions: Dietary Supplement: Postbiotic
- Placebo (Placebo Comparator): Arm receiving placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Postbiotic — multistrain postbiotic in the form of a capsule with a daily dose of 1E+9 Colony Forming Unit (CFU) per day for 6 weeks.
  Arms: Active
Dietary Supplement: Placebo — Matching placebo in a form of a capsule for 6 weeks.
  Arms: Placebo

SUMMARY:
This study evaluates the efficacy of a multistrain postbiotic administered in the form of a capsule in the management of moderate self-reported anxiety in adults aged 18-65

DETAILED DESCRIPTION:
The subjects will be placebo non-responders from part 1 of the trial, looking at the effect of a multistrain probiotic on anxiety.

ELIGIBILITY:
Inclusion Criteria:

1. Be able to give written informed consent.
2. Be between 18 to 65 years inclusive.
3. Mild to moderate self-reported anxiety
4. Have a Beck Depression Inventory (BDI) score <20.
5. Is in general good health, as determined by the investigator.
6. Be willing to maintain stable dietary habits and physical activity levels throughout the study period.
7. Be able to communicate well with the Investigator, to understand and comply with the requirements of the study and be judged suitable for the study in the opinion of the Investigator.
8. Willing to consume the study product daily for the duration of the trial and comply with all trial procedures.
9. Be able to give confirmation of ongoing informed consent from Part 1 of the trial.
10. Has been allocated to the placebo arm of Part I of the trial
11. Has been deemed a "non-responder" in Part I of the trial

Exclusion Criteria:

1. Are less than 18 or greater than 65.
2. Participants who are pregnant or wish to become pregnant during the trial.
3. Participants who are lactating and/or currently breastfeeding
4. Participants currently of childbearing potential, but not using an effective method of contraception, as outlined below:
5. Complete abstinence from intercourse two weeks prior to administration of the study product, throughout the clinical trial, until the completion of follow-up procedures or for two weeks following discontinuation of the study product in cases where Participant discontinues the trial prematurely. (Participants utilising this method must agree to use an alternate method of contraception if they should become sexually active and will be queried on whether they have been abstinent in the preceding 2 weeks when they present to the clinic for the Final Visit).
6. Has a male sexual partner who is surgically sterilised prior to the Screening Visit and is the only male sexual partner for that Participant.
7. Sexual partner(s) is/are exclusively female.
8. Use of acceptable method of contraception, such as a spermicide, mechanical barrier (e.g. male condom, female diaphragm), tubal ligation or contraceptive pill. The Participant must be using this method for at least 1 week prior to and 1 week following the end of the trial.
9. Use of any intrauterine device (IUD) or contraceptive implant. The Participant must have the device inserted at least 2 weeks prior to the first Screening Visit, throughout the trial, and 2 weeks following the end of the trial.
10. Are hypersensitive to any of the components of the study product.
11. Has taken systemic antibiotics within the previous 8 weeks.
12. Has taken probiotics or post-biotics within the previous 8 weeks.
13. Has a current clinical diagnosis of depression - determined in their medical history.
14. Has self-reported or suspected consumption of excess quantities of alcohol or recreational drugs
15. Diagnosed with significant physical comorbidity that, in the investigator's judgment, precludes involvement in the study.
16. Has an acute or chronic illness (e.g., heart disease, inflammatory bowel disease, cancer, HIV) that, in the Investigators judgment, precludes involvement in the study.
17. Participants who have received cognitive behavioural therapy (CBT) or psychotherapy in the 8 weeks prior to baseline or plan to start during the period of the study.
18. Participants who have taken anti-depressants or supplements known to impact mood (e.g., valerian, St. John's Wort) in the 8 weeks prior to baseline or planning to start in the study period.
19. Taking dietary supplements or food products that the investigator believes would interfere with the objectives of the study within 8 weeks prior to baseline ;
20. Participants who have taken psychotropics, anxiolytics, antipsychotics, anticonvulsants, systemic corticosteroids, opioid pain relievers, hypnotics, and/or prescribed sleep medication within 8-weeks of screening.
21. Has a gastrointestinal disease or condition, that by the investigators judgement, could interfere with the intestinal barrier function.
22. Are severely immunocompromised (transplant patient, on antirejection medications, on a steroid for 30 days, or chemotherapy or radiotherapy within the last year; HIV positive participants with undetectable viral loads would be allowed on the trial)
23. Have an active malignant disease or any concomitant end-stage organ disease (in the last 12 months), which, in the Investigator's judgment, contraindicates participation in the study.
24. Any immunosuppressant or chemotherapy medications, including mercaptopurine, azathioprine, or methotrexate;
25. Have had any other condition or are taking a medication that the investigator believes would interfere with the objectives of the study, pose a safety risk, or confound the interpretation of the study results
26. Individuals who, in the opinion of the investigator, are considered to be poor attendees or unlikely for any reason to be able to comply with the trial.
27. Participants may not be receiving treatment involving experimental drugs. If the Participant has been in a recent experimental trial, these must have been completed not less than 8 weeks prior to this trial.
28. Any Participant who is an employee of the study site or an Atlantia Clinical Trials employee or their close family member or a member of their household.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-01-04 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Change in Anxiety rating | Day 0, Day 42
  Level of anxiety measured with "Hamilton Anxiety Rating Scale". (max 56 points) where a lower score means better outcomes compared to baseline.

SECONDARY OUTCOMES:
Change in Depression score | Day 0, Day 42
  Level of depression measured with "Beck's Depression Inventory". (max 63 points) where a lower score means better outcomes compared to baseline.
Change in Depression score | Day 0, Day 42
  Level of depression measured with "Patient Health Questionnaire 9". (max 27 points) where a lower score means better outcomes compared to baseline.
Change in trait anxiety | Day 0, Day 42
  Level of trait anxiety measured with "State-Trait Anxiety Inventory" (max 80 points) where a lower score means better outcomes compared to baseline.
Change in perceived stress | Day 0, Day 42
  Level of perceived stress measured with "Cohen's perceived Stress scale" (max 40 points ) where a lower score means better outcomes compared to baseline.
Change in Stress | Day 0, Day 42
  Level of stress measured with "Salivary Cortisol awakening response" (ng/dL).
Change in Sleep Quality | Day 0, Day 42
  Change in sleep quality measured by "Pittsburgh Sleep Quality Index" (max 21 points) where a lower score means better outcomes compared to baseline.
Change in Gastrotintestinal symptoms | Day 0, Day 42
  Degree of GI symptoms measured by "GI Symptom Rating Scale" where a lower score means better outcomes compared to baseline.
Change in Quality of Life evaluation | Day 0, Day 42
  Change in quality of life score measured by the "SF-36 questionnaire" (max 100 points) where a higher score means better outcomes compared to baseline.

OTHER OUTCOMES:
Change in GI microbiome | Day 0, Day 42
  Faecal microbiome analysis assessed by metagenomics.

CONTACTS AND LOCATIONS:
Locations (1):
- Atlantia Food Clinical Trials, Cork, Ireland

IPD SHARING:
Plan to Share IPD: No